3D Breast Imaging for Cosmetic and Reconstructive Breast Surgery: Does 3D Improve Patient Reported Outcomes in Primary Breast Augmentation?

NCT01964105

AUGUST 27, 2014

The trend of enrolling to the randomized arm of our study will be modeled using the LOGISTIC procedure with maximum likelihood estimation. Predicted probability will be obtained from this model to facilitate clear interpretation of non-linear relationships with time. For patient-level comparisons, the assumption of normality will be examined with the Shapiro-Wilk test after which a t-test or Wilcoxon test will be used as appropriate. When using the t-test, equality of variances will first be examined with the Folded F statistic. The pooled t-test will be used for two populations with equal variances. Otherwise the Satterthwaite t-test will be used. Breast-level comparisons will be performed using generalized estimating equations (GEE) and empirical standard error estimates to account for correlation of left and right breast measurements within the same patient. The Pearson or Spearman correlation coefficient will be used to quantify the direction and magnitude of association between mammometric, Q-Score, and clinical data. Statistical analyses will be performed in SAS, version 9.4, with descriptive statistics analyzed and graphed in Prism 7 for Mac.